CLINICAL TRIAL: NCT02755922
Title: Bone Regeneration in Mandibular Fractures After the Application of Autologous Mesenchymal Stem Cells. Randomized Clinical Trial.
Brief Title: Bone Regeneration With Mesenchymal Stem Cells
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Alejandro Gonzalez-Ojeda, M.D.,Ph.D., F.A.C.S., Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-1301-27
Record Dates: First submitted 2016-04-20; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Mandibular Fractures
Keywords: Mesenchymal Stem Cells; Treatment
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fractures with Mesenchymal Stem Cells (Experimental): 10 patients with mandibular fractures were managed by open reduction and internal fixation, with application of autologous mesenchymal stem cells on the fracture site.
  Interventions: Biological: Application of autologous mesenchymal stem cells
- Fractures without Mesenchymal Stem Cells (No Intervention): 10 patients with mandibular fractures were managed by open reduction and internal fixation, without application of autologous mesenchymal stem cells on the fracture site.

INTERVENTIONS:
Biological: Application of autologous mesenchymal stem cells — within the surgical procedure, mesenchymal stem cells, were applied on the fracture site. Imaging by X-ray and CT and imaging analysis was done after fracture repair, at week 4 and week 12
  Arms: Fractures with Mesenchymal Stem Cells

SUMMARY:
Mandible fractures are a common cause of facial injury in adults. The autologous mesenchymal stem cell (AMSC) transplantation, is proposed as an alternative to the conventional graft treatment, improving bone neoformation.The objective was to evaluate the effectiveness of AMSCs application in mandibular fractures to reduce regeneration time and increase bone quality.

DETAILED DESCRIPTION:
Single blinded controlled clinical trial in patients with mandibular angle fracture. The patients were divided into: Study Group (SG): fracture reduction plus application of AMSCs, Control Group (CG): Same procedure without AMSCs. AMSCs were obtained from adipose tissue , 24 hrs before the procedure. Intensity and density were evaluated in normal bone and fractured bone, at 4 and 12 weeks after surgery using panoramic radiography and computed tomography. (CT)

A total of 20 patients, 10 in each group were included. SG with a mean age of 31.2 ± 6.3 years and CG 29.7 ± 7.2 years, all patients were male. Bone quality at week 4 SG 108.82 ± 3.4 vs CG 93.92 ± 2.6 (p = 0.000) by panoramic radiography, SG 123 ± 4.53 vs CG 99.72 ± 5.72 (p = 0.000) by CT. At week 12: SG 153.53±1.83 vs CG 101.81±4.83 (p= 0.000) by panoramic radiography, SG 165.4 ± 4.2 vs CG 112.05±2.1 (p= 0.000) by CT.

The application of AMSCs presented at week 4 similar ossification values compared with normal bone and a 36.48 % higher ossification rate at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Entitled patients to the Mexican Institute of Social Security
* Patients with mandibular condyle fractures associated or not to other initial fracture that required Open reduction and internal fixation
* Ages from 17 to 59 years
* Both female and male gender
* Patients who gave their consent to be part of this trial

Exclusion Criteria:

* Patients younger than 17 years and older than 59 years
* Chronic-degenerative diseases, active smoking, collagen disorders
* Patients with signs of infection in the aimed area to treat and in whom the fracture occurred in a longer period than 10 days before their surgery.

Ages: 17 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change of bone quality | from the moment of fracture diagnosis to week 4 and week 12 after surgery
  After the procedure, imaging control by X-ray and analysis by software, was done after surgery at weeks 4 and 12. X- ray units: Voxels. Software analysis by Image Processing and Analysis ImageJ 1.43
Change of bone quality | from the moment of fracture diagnosis to week 4 and week 12 after surgery
  After the procedure, imaging control by CT scan and analysis by software, was done after surgery at weeks 4 and 12. CT scan units: Hounsfiled . Software analysis by Image Processing and Analysis ImageJ 1.43

SECONDARY OUTCOMES:
Number of patients with infection ( increase of local temperature, tenderness, leukocyte count >10,000/ µL, confirmed by Gram stain and blood culture). | from immediate postoperative period to three months after surgery
  Infection suggested by clinical diagnosis increase of leukocyte levels, and confirmed by Gram stain and blood culture of local sample.
Number of patients with bleeding after surgery (Persistent bleeding, ineffectiveness stopping bleeding using dressings) | from immediate postoperative period to 1 week after surgery
  Persistent bleeding after surgery, that did not stop by dressings. If this complication developed, it had to be managed by surgical techniques.
Number of patients with surgical wound dehiscence (subcutaneous tissue , bone or osteosynthesis material exposed and seen through opened skin ) | from immediate postoperative period to one month
  Clinical signs of dehiscence on the surgical incision, surgical material or bone seen though the skin. This diagnosis is done by clinical findings. Does not need any laboratory or image test.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gonzalez Ojeda, M.D., Ph.D., Principal Investigator — Instituto Mexicano del Seguro Social

IPD SHARING:
Plan to Share IPD: Yes